CLINICAL TRIAL: NCT05844865
Title: Patient Derived Vascularized MicroTumor Model of Gastrointestinal Peritoneal Carcinomatosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Maheswari Senthil, MD, Professor of Surgery, Division Chief - Surgical Oncology, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2214; UCI 22-92 (Other: CFCCC)
Record Dates: First submitted 2023-01-27; First posted 2023-05-06 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Peritoneal Carcinomatosis; Gastrointestinal Peritoneal Carcinomatosis
Keywords: Peritoneal Carcinomatosis; Gastrointestinal Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects with Gastrointestinal Primary Tumor with or without Peritoneal Carcinomatosis (Other): Subjects with gastrointestinal (GI) primary tumor with or without peritoneal carcinomatosis who are undergoing planned standard of care (SOC) surgical procedures. Biospecimens such as blood, peritoneal wash fluid and tumor samples will be obtained.
  Interventions: Other: Biospecimen Collection (Blood, Ascites/Peritoneal Wash Fluid and/or Tumor Samples)

INTERVENTIONS:
Other: Biospecimen Collection (Blood, Ascites/Peritoneal Wash Fluid and/or Tumor Samples) — Subjects with a known diagnosis of GI primary tumor with or without PC, with a planned standard of care surgery.

SUMMARY:
This is a pilot study gathering and using samples and data from patients with gastrointestinal peritoneal carcinomatosis. Participants will be asked for permission to provide blood and ascites/peritoneal wash fluid, tumor samples during their planned surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a GI tumor
* Must have planned standard of care surgical procedure
* Age ≥ 18 years.
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

- Pattens who are unable to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Establishment of angioarchitechture of peritoneal lesions through Optical Coherence Tomography Angiography (OCTA) | Up to 4 years
  Establishment and evaluation of angioarchitecture of peritoneal lesions through OCTA imaging obtained during surgery.
Development of individual patient-derived peritoneal carcinomatosis (pdPC) vascularized micro-tumor (VMT) | Up to 4 years
  Successful establishment of multicellular pdPC VMT models from metastatic and/or primary tumor tissue with increasing tumor volume over a 14 day period.

SECONDARY OUTCOMES:
Compare response of therapeutic regimens in a pdPC VMT to the observed clinical response (by RECIST criteria or diagnostic laparoscopy) | Up to 4 years
  Response to therapy in a pdPC VMT will be correlated with the clinical response observed in patients treated with similar regimens using either RECIST criteria if measurable disease is available or by diagnostic laparoscopy performed as part of standard of care to assess treatment response
Progression-Free Survival (PFS) at 6 months | 6 months
  Survival analysis will utilized to study association between in vitro model and patient clinical response. Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Estimates at 6 months will be made.
Overall Survival (OS) | Up to 4 years
  Survival analysis will utilized to study association between in vitro model and patient clinical response. The duration of time from start of treatment to time of progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Maheswari Senthil, MD FACS, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States